CLINICAL TRIAL: NCT03406273
Title: A Standardized Protocol of Surgery and Radiation for Patients With Brain Metastases in Relapsed Neuroblastoma
Brief Title: Standardized Protocol of Surgery and Radiation for Patients With Brain Metastases in Relapsed Neuroblastoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment to study, study closed
Sponsor: Giselle Sholler (Other)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Beat Childhood Cancer Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HITC001
Record Dates: First submitted 2018-01-08; First posted 2018-01-23 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Relapsed Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Radiation; Spermine Synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ≥ 5 years of age (Experimental): Cerebral Spinal (CS) radiation
  Interventions: Radiation: Cerebral Spinal (CS) radiation
- < 5 yo and ≥ 3 yo and CSF + (Experimental): Cerebral Spinal (CS) radiation
  Interventions: Radiation: Cerebral Spinal (CS) radiation
- All < 3 yo & < 5 yo/≥ 3 yo CSF neg (Experimental): Focal radiotherapy (SRS)
  Interventions: Radiation: Focal radiotherapy (SRS)

INTERVENTIONS:
Radiation: Cerebral Spinal (CS) radiation — Surgery plus Cerebral Spinal (CS) radiation
  Arms: < 5 yo and ≥ 3 yo and CSF +; ≥ 5 years of age
Radiation: Focal radiotherapy (SRS) — Surgery plus focal radiotherapy (stereotactic radiosurgery to the tumor bed [SRS])
  Arms: All < 3 yo & < 5 yo/≥ 3 yo CSF neg

SUMMARY:
HITC001 is a single institution study to evaluate the efficacy of using a standardized protocol of surgery and radiation for patients with brain metastases in relapsed neuroblastoma.

DETAILED DESCRIPTION:
This clinical trial aims to establish a standardized protocol consisting of surgery and radiation for patients with brain metastases in relapsed neuroblastoma. This will be an adjunct study to NMTRC009 onto which patients will be enrolled to for treatment with precision therapy. This study will follow the efficacy, safety, and CNS progression-free survival of surgery and radiation.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≤ 21 years at the time of study entry.
* Diagnosis: Histologic verification at either the time of original diagnosis or relapse of neuroblastoma.
* Disease Status: Patients must have ONE of the following along with disease in the CNS:

  1. Any episode of recurrent disease following completion of aggressive multi-drug frontline therapy.
  2. Any episode of progressive disease during aggressive multi-drug frontline therapy.
  3. Primary resistant/refractory disease detected at the conclusion of at least 4 cycles of aggressive multidrug induction chemotherapy on or according to a high-risk neuroblastoma protocols.
* Measurable or evaluable disease by Brain MRI.
* Current disease state must be one for which there is currently no known curative therapy.
* Meet all inclusion criteria for study NMTRC009
* Informed Consent: All subjects and/or legal guardians must sign informed written consent. Assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Meets all exclusion criteria for study NMTRC009
* Subjects who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study, or in whom compliance is likely to be suboptimal, should be excluded.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05 (Estimated); Primary Completion 2017-05-01 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) of Participants by the presence of radiologically measurable CNS disease by cross-sectional CT or MRI imaging and/or by MIBG or PET scans and/or CSF Sampling. | 3 years
  To determine the activity of treatments chosen based on Overall response rate (ORR) using RESIST criteria.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety | 3 years
  To determine the safety of using a standardized protocol of surgery and radiation for patients with brain metastases in relapse neuroblastoma
Progression Free Survival (PFS) interval for CNS lesions will be measured by days from start of treatment (surgery/radiation) to the date of any future progressive disease (PD) in CNS lesions per RESIST criteria. | 3 years
  Time to progression (PFS), defined as the period from the start of the treatment until the criteria for progression are met taking as reference the screening measurements
Length of time that participants experience Overall Survival (OS) | 8 years
  Overall survival (OS) will be defined as the period in days from the date of enrollment until the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Kaveh Asadi-Moghaddam, MD, Study Chair — Corewell Health West
Locations (1):
- Helen DeVos Children's Hospital, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No